CLINICAL TRIAL: NCT04484402
Title: Treatment of Patients With Inflammatory-dystrophic Diseases of the Cornea Using Autologous Limbal Stem Cells (Corneal Epithelial Stem Cells) or Adipose-derived Mesenchymal Stem Cells
Brief Title: Treatment of Patients With Inflammatory-dystrophic Diseases of the Cornea Using Autologous Stem Cells
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus (Other Government)
Collaborators: Belarusian State Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBCE_LSC
Record Dates: First submitted 2020-07-20; First posted 2020-07-23 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Corneal Ulcer; Corneal Disease; Corneal Dystrophy
Keywords: Corneal Disease
MeSH Terms: conditions — Corneal Ulcer; Corneal Diseases; Corneal Dystrophies, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- mesenchymal stem cells (Experimental): Patients with inflammatory-dystrophic diseases of the cornea receiving standard treatment plus adipose-derived mesenchymal stem cells
  Interventions: Biological: mesenchymal stem cells; Other: standard treatment
- limbal stem cells (Experimental): Patients with inflammatory-dystrophic diseases of the cornea receiving standard treatment plus adipose-derived limbal stem cells
  Interventions: Biological: limbal stem cells; Other: standard treatment
- control (Active Comparator): Patients with inflammatory-dystrophic diseases of the cornea receiving standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Biological: mesenchymal stem cells — Autologous adipose-derived mesenchymal stem cells mixed with sodium hyaluronate 1% solution
  Arms: mesenchymal stem cells
Biological: limbal stem cells — Autologous adipose-derived limbal stem cells mixed with sodium hyaluronate 1% solution
  Arms: limbal stem cells
Other: standard treatment — Standard treatment according to the Clinical protocols

SUMMARY:
Treatment of patients with inflammatory-dystrophic diseases of the cornea using autologous limbal stem cells (corneal epithelial stem cells) or adipose-derived mesenchymal stem cells

DETAILED DESCRIPTION:
In order to treat inflammatory and dystrophic diseases of the cornea perilimbal injections of cultured autologous stem cells are performed. Corneal (limbal) epithelial stem cells (LSC) or mesenchymal stem cells derived from adipose tissue (ADSC) are mixed with sodium hyaluronate 1%

ELIGIBILITY:
Inclusion Criteria:

* inflammatory-dystrophic diseases of the cornea:

  1. Epithelial defects of the cornea, ulcerative keratitis of various etiology, resistant to standard methods of treatment
  2. Dystrophic diseases of the cornea, accompanied by edema
  3. Burns of the cornea
  4. Neurotrophic forms of keratitis
  5. Persistent post-traumatic, postoperative, contusion keratitis and keratopathy

Exclusion Criteria:

1. Pregnancy.
2. Viral hepatitis B and C, HIV, tubeculosis and other chronic viral and bacterial infections.
3. Cancer or leukemia
4. Any diseases in the stage of decompensation.
5. Mental disorders.
6. Anomalies of eye refraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Number of cured patients | 2 month
  Number of patients cured
Number of patients with treatment-related adverse events | 4 weeks
  MSC/LSC application related adverse events assessed by blood count, liver and function tests

CONTACTS AND LOCATIONS:
Overall Officials: Igor Volotovski, Prof, Study Director — Head of the Lab of Institute of Biophysics and Cell Engineering; Liudmila Marchenko, Prof, Study Director — Head of the Department of eyes diseases of Belarusian State Medical University; Zinaida Kvacheva, Principal Investigator — Leading researcher, Institute of Biophysics and Cell Engineering
Locations (1):
- Institute of Biophysics and Cell Engineering of National Academy of Sciences of Belarus, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: No